CLINICAL TRIAL: NCT05411497
Title: Use of Natural Signals and Ambient Dendritic Cells to Culture-Expand Cancer Targeting T-Cells Directly From Unfractionated Peripheral Blood: A Phase 1 T-Cell Dose Escalation Trial Targeting Relapsed and Refractory MUC1-Expressing Multiple Myeloma
Brief Title: Genetically Engineered Cells (MUC1-Activated T-Cells) for the Treatment of MUC1 Positive Recurrent or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200806; NCI-2022-03111 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-001202 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-06-09 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, MUC1-activated T-cells) (Experimental): LD CHEMOTHERAPY: Patients receive cyclophosphamide IV over 60 minutes on days -5, -4, -3.
  ASCT: Patients receive MUC1-activated T-cells IV over 10 minutes to 1 hour on day 0.
  Interventions: Biological: Autologous MUC1-activated T-cells; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Autologous MUC1-activated T-cells — Given IV
  Other Names: Autologous MUC1-activated T-lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719

SUMMARY:
This phase I trial tests the safety, side effects and best dose of MUC1-activated T cells in treating patients with multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory) and is positive for expression of the MUC1 protein. T-cells are infection fighting blood cells that can kill cancer cells. MUC1-activated T-cells are made from the body's own T cells. The manufactured T-cells are made to target the MUC1 genetic marker and may help the body's immune system identify and kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the toxicity of in-house, manufactured MUC1-activated T cells in patients with relapsed/refractory MUC1-expressing multiple myeloma.

SECONDARY OBJECTIVES:

I. Obtain preliminary efficacy associated with MUC1-targeting peripheral blood mononuclear cells (PBMC) derived T cells in conjunction with cyclophosphamide (CTX) in MUC1-expressing multiple myeloma patients.

Ia. Assess best objective response observed based on International Myeloma Working Group (IMWG) criteria and duration of any partial or complete responses (partial response [PR] or complete response [CR]).

Ib. Assess progression-free (PFS) and overall (OS) survival. II. Determine feasibility of production and administration of MUC1-targeting PBMC-derived T cells and ability to proceed with T cell dose escalation.

IIa. Assess the feasibility of in-house preparation of in vitro-sensitized T cells.

III. Evaluate the safety, including all grades of neurotoxicity immune effector cell associated neurotoxicity (ICANS) and cytokine release syndrome (CRS) as determined by American Society of Transplantation and Cell Therapy (ASTCT) criteria, by monitoring adverse events, laboratory abnormalities, vital signs, and other safety parameters.

IV. Estimate the incidence of Grade 3 or higher of neurotoxicity and cytokine release syndrome by Grade 3 or higher neurotoxicity (ICANS) or CRS per the ASTCT criteria.

V. Assess efficacy of a single dose of MUC1-activated T cells.

CORRELATIVE RESEARCH OBJECTIVES:

I. Perform analyses of Vbeta usage by T cell receptors (TCR) to see whether culture expansion generated TCR oligoclonality; whether such T cells persist in the circulation following adoptive transfer; and whether such persistence significantly correlates to objective responses.

Ia. Levels of Vbeta alleles on CD3+ T cells in blood by antibody staining or deoxyribonucleic acid (DNA) sequencing (Adaptive Biotechnologies).

II. Characterize the changes in cytokine levels over time. III. Determine whether T cells recognizing MUC1 in an major histocompatibility complex (MHC)-restricted manner in culture (intracellular IFN-gamma assays) correspond to therapeutic efficacy upon subsequent adoptive transfer.

IV. Determine the immune phenotype of the immune cells, the inhibitory profile, and transcription factors using multi-color flow cytometry.

V. Assess hospital resource utilization and health economics.

OUTLINE: This is a dose-escalation study of MUC1-activated T-cells.

LYMPHODEPLETION (LD) CHEMOTHERAPY : Patients receive cyclophosphamide intravenously (IV) over 60 minutes on days -5, -4, -3.

AUTOLOGOUS STEM CELL TRANSPLANTATION (ASCT): Patients receive MUC1-activated T-cells IV over 10 minutes to 1 hour on day 0.

After completion of study treatment, patients are followed up on days 1, 2, 3, 7, 28 and every 90 days for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* MUC1 expression in multiple myeloma tumor cells verified by immunohistochemistry (IHC) or flow cytometry (FCM). Heterogeneous tumor expression of MUC1 is acceptable
* Relapsed or refractory multiple myeloma previously treated with or intolerant to at least three prior lines of therapy and be relapsed or intolerant to a proteasome inhibitor, an immune modulatory drug (IMiD), and a CD38 antibody. Patients must be at least 90 days since an autologous stem cell transplant, if performed
* Patients must have measurable disease per IMWG criteria on study entry, which must include at least one of the following:

  * Serum M-spike >= 0.5 g/dL Patients with IgA, IgM or IgD myeloma in whom serum protein electrophoresis is deemed unreliable for routine M-protein quantitation may be considered eligible if total serum IgA, IgM or IgD level is elevated above normal range and parallels disease course
  * 24-hour urine M-spike >= 200 mg
  * Involved serum free light chain (FLC) >= 10 mg/L with an abnormal free light chain ratio
  * Bone marrow plasma cells > 30%
  * Patients with extramedullary disease:

    * 1 lesion that has a single diameter of >= 2 cm measured by computed tomography (CT) or magnetic resonance imaging (MRI) or the CT portion of the positron emission tomography (PET)/CT
    * Skin lesions can be used if the area is >= 2cm in at least one diameter and measured with a ruler
* Willingness and ability to provide written informed consent
* Willing to return to Mayo Clinic Hospital in Arizona (MCA) for follow-up during the active monitoring phase of the study
* Willingness to provide mandatory blood, bone marrow biopsy, and aspirate specimens for correlative research
* Willing to undergo leukapheresis for blood component collection
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 14 days of study registration)
* Lymphocyte count >= 500/mm^3 (within 14 days of study registration)
* Hemoglobin >= 8.0 g/dL (within 14 days of study registration)
* Platelet count >= 30,000/mm^3 (within 14 days of study registration)
* Total bilirubin =< 2.0 mg/dL unless patient has documented Gilbert's syndrome (Subjects with Gilbert's Syndrome may be included if their total Bilirubin is =< 3.0 x upper limit of normal (ULN) and direct bilirubin =< 1.5 x ULN) (within 14 days of study registration)
* Alanine aminotransferase (ALT) and aspartate amino transferase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement of their cancer) (within 14 days of study registration)
* Prothrombin time, international normalized ratio (PT, INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulation therapy and INR or aPTT is within target range of therapy (for patients receiving anticoagulation, there should be no prior history of bleeding and no recent deep vein thrombosis [DVT]/pulmonary embolism [PE] within the last 6 months of enrollment)
* Calculated creatinine clearance >= 30 ml/min using the Cockcroft-Gault formula (within 14 days of study registration)
* Baseline oxygen saturation >= 90% on room air

Exclusion Criteria:

* Clinically unresolved central nervous system (CNS) metastases
* Prior treatment targeting MUC1
* Subjects with known plasma cell leukemia (PCL)
* Any of the following are excluded because this study involves an agent (CTX) that has known genotoxic, mutagenic and/or teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate birth control measures
* History of myocardial infarction >= 6 months prior to registration, and/or congestive heart failure requiring ongoing treatment such as medications and/or an implanted defibrillator to control life-threatening arrhythmias.
* Failure to recover to grade 1 or baseline from acute, reversible effects of prior therapy regardless of interval since last treatment.

EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment.

* Uncontrolled concurrent illness including, but not limited to:

  * Inability to clear an ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled psychiatric problems and/or difficult social situation
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that the protocol investigators deem could potentially limit compliance with study requirements
* Evidence of clinical immunocompromise and/or human immunodeficiency virus (HIV) positivity and currently receiving antiretroviral therapy
* Patients requiring chronic supraphysiologic daily doses of steroids (>10 mg prednisone or prednisolone, >= 4 mg Decadron or >= 50 mg hydrocortisol daily)
* Patients receiving any other investigational agent which could be considered a treatment for the neoplasm
* Other active malignancy first documented =< 4 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history of other malignancy, the patient must not be receiving other treatment aimed at suppressing its recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2027-08-18 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 4 years

SECONDARY OUTCOMES:
Clinical response | Up to 4 years
  The number of responses (complete response [CR], very good partial response [VGPR], partial response [PR], or minimal response [MR]) will be summarized by simple descriptive summary statistics. Assuming that the number of responses is binomially distributed, we will estimate the proportion of patients who achieve an overall as well as specific type of response along with corresponding 95% exact binomial confidence intervals.
Progression-free survival | From registration to disease progression or death due to any cause, assessed up to 4 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (overall and by dose level). Given the nature of phase I trials and the limited numbers, this endpoint will be primarily descriptive and to characterize the patients enrolled.
Overall survival | From registration to death due to any cause, assessed up to 4 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier (overall and by dose level).

OTHER OUTCOMES:
Pharmacodynamics, adoptive T cells immunophenotyping TCRVbeta | Up to 4 years
  Whole blood will be collected sent to the Hematologic Malignancies Laboratory for TCR Vbeta repertoire of the T cells and phenotypes and ex vivo functions prior to infusion and 1 day after the infusion, 1 week later, and one month later and then every 3 months for two years. This testing will also be performed on the leukapheresis product. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).
Pharmacodynamics, immune cell profiling (whole blood) | Up to 4 years
  Whole blood will be collected at the indicated time points and sent to the Hematologic Malignancies Laboratory. Assessment of immune response will be done in Human Cell Therapy Laboratory. Depending on preliminary results, future analysis may not proceed. This testing will also be performed on the leukapheresis product. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).
Pharmacodynamics, cytokines (plasma) | Up to 4 years
  Whole blood will be collected and sent to the Hematologic Malignancies Laboratory for plasma isolation processing and initial cryopreservation. Analyses will be batched. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).
Pharmacodynamics, immune and tumor and phenotype (bone marrow) | Up to 4 years
  Whole bone marrow aspirate will be collected and sent to the Hematologic Malignancies lab for immune cell profiling. Central vendor, Adaptive Biotech, will provide shipping supplies. Sample shipping and analysis will be done in batches. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).
MUC1 expression (bone marrow biopsy tissue/slides) | Up to 4 years
  Slides will be made, via retrospective request, from bone marrow biopsy tissue stored in Hematopathology clinical archives. Micron thickness should be 5um. Central vendor NeoGenomics will provide kits, shipping supplies and pre-paid shipping labels. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).
MUC1 expression (bone marrow aspirate) | Up to 4 years
  Whole bone marrow aspirate will be collected and sent to the Hematologic Malignancies lab for FCM. If there is no detectable MUC1 staining other correlative studies will not be performed and the patient will go off study. Descriptive statistics and scatterplots will form the basis of presentation of these variables. Correlations between the laboratory values and other outcome measures will be carried out by standard parametric and non-parametric tests (e.g., Pearson's and Spearman's rho).

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergsagel, M.D., Principal Investigator — Mayo Clinic Hospital in Arizona
Locations (2):
- United States (2):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials